CLINICAL TRIAL: NCT06239038
Title: Does Electrocautery Increase Postoperative Pain in Primary Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Does Electrocautery Increase Postoperative Pain in Primary Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Police General Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Pawut Wattanapongsiri, Principal investigator, Police General Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGH protocal
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee arthroplasty, Electrocautery, Scalpel, Post-operative pain, Pain score
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: In electrocautery group, using an electrocautery in following step
  1. Stop bleeding at subcutaneous tissue layer
  2. Remove anterior cruciate ligament and posterior cruciate ligament
  3. Bony mark for further bone cut
  4. Patellar denervation
  5. Soft tissue removal
  6. Synovial tissue removal
  In scalpel group, proceed with following step
  1. Using electrocautery for stop bleeding at subcutaneous tissue layer
  2. In deep layer still use scalpel for Remove anterior cruciate ligament and posterior cruciate ligament
  3. Soft tissue removal and synovial tissue removal
  4. No patellar denervation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scalpel group (Experimental): Proceed with following step
  1. Using electrocautery for stop bleeding at subcutaneous tissue layer
  2. In deep layer still use scalpel for Remove anterior cruciate ligament and posterior cruciate ligament
  3. Soft tissue removal and synovial tissue removal
  4. No patellar denervation
  Interventions: Procedure: total knee arthroplasty
- electrocautery group (Experimental): Using an electrocautery in following step
  1. Stop bleeding at subcutaneous tissue layer
  2. Remove anterior cruciate ligament and posterior cruciate ligament
  3. Bony mark for further bone cut
  4. Patellar denervation
  5. Soft tissue removal
  6. Synovial tissue removal
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — total knee arthroplasty surgery with Police Arthroplasty joint academy center(PAJAC) Subvastus Approach

SUMMARY:
Total knee arthroplasty (TKA) is a successful treatment for end-stage osteoarthritis of the knee. The main advantages of TKA are to relieve the pain of the knee, improve the knee function, restore lower limb alignment, and improve the quality of life for patients. During TKA, some surgeons prefer using a scalpel while others using electrocautery to expose the articular cavity. Whether the use of scalpel can lead to better and faster recovery after the primary TKA is still controversial.

The aim of this study was to compare the clinical outcomes of using the scalpel and the electrocautery in primary TKA

DETAILED DESCRIPTION:
A randomized controlled trial of patients underwent primary TKA between October 2021 and October 2023. The groups will be determined by using the computer to generate a randomization lists. A total 132 patients were included with 66 patients in the scalpel group, 66 patients in the electrocautery group. All patients were evaluated using primary outcome : Post-operative Visual Analog Scale (VAS) of pain, secondary outcome: estimated blood loss and Knee Injury and Osteoarthritis Outcome Score (KOOS-JR)

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis patient (KL classification gr 2-4)
* Primary TKA
* Varus deformity < 20 degree
* Flexion contracture < 20 degree

Exclusion Criteria:

* Coagulopathy
* Platelet dysfunction
* Inflammatory arthritis
* Revision TKA

Min Age: 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain (visual analog scale) day 1-4 | postoperative day 1-4
  measure the Postoperative pain by using visual analog scale from 1 - 10, higher scores means worse outcome

SECONDARY OUTCOMES:
Calculated blood loss | postoperative day 4
  Calculated blood loss using Mercuruali's formula
Functional score | follow up 2 weeks, 1,3,6 months
  Functional score using KOOS JR score, range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health

CONTACTS AND LOCATIONS:
Overall Officials: Pawut Wattanapongsiri, Principal Investigator — orthopedic department, Police General Hospital, Thailand
Locations (1):
- Police General Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No